CLINICAL TRIAL: NCT03910530
Title: A Phase 1b Study of INCMGA00012 (PD-1 Inhibitor), INCB001158 (Arginase Inhibitor), and the Combination in Japanese Participants With Advanced Solid Tumors
Brief Title: A Study of INCMGA00012, INCB001158, and the Combination in Japanese Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCMGA 0012-104
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Advanced solid tumors; metastatic solid tumors; INCMGA00012; INCB001158; Japan; PD-1 Inhibitor; Arginase Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- INCMGA00012 (Experimental): Single-agent INCMGA00012.
  Interventions: Drug: Retifanlimab
- INCB001158 75 mg (Experimental): Single-agent INCB001158.
  Interventions: Drug: INCB001158
- INCB001158 100 mg (Experimental): Single-agent INCB001158.
  Interventions: Drug: INCB001158
- INCMGA00012 + INCB001158 (Experimental): Combination of INCMGA00012 and INCB001158.
  Interventions: Drug: Retifanlimab + INCB001158

INTERVENTIONS:
Drug: Retifanlimab — Part 1: INCMGA00012 500 mg every 4 weeks administered intravenously over 60 minutes.
  Other Names: INCMGA00012
  Arms: INCMGA00012
Drug: INCB001158 — Part 1: INCB001158 75 or 100 mg twice daily administered orally.
  Arms: INCB001158 100 mg; INCB001158 75 mg
Drug: Retifanlimab + INCB001158 — Part 2: INCB001158 at the recommended Phase 2 dose selected from Part 1 in combination with INCMGA00012 .
  Other Names: INCMGA00012
  Arms: INCMGA00012 + INCB001158

SUMMARY:
The purpose of this study is to assess the safety and tolerability and the pharmacokinetics (PK) of INCMGA00012 (PD-1 Inhibitor), INCB001158 (Arginase Inhibitor), and the combination in Japanese participants with advanced solid tumor malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Participant is Japanese
* Histologically or cytologically confirmed diagnosis of any locally advanced or metastatic solid tumors not amenable to local or other curative therapy.
* Participants with nonevaluable lesions are allowed.
* Life expectancy > 3 months.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Female participants agree to use medically acceptable contraceptive measures, should not be breastfeeding, and must have a negative pregnancy test before the start of study drug administration.
* Female participants of childbearing potential must understand and accept that pregnancy must be avoided during participation in the study.
* Male participants should avoid unprotected sex with women of childbearing potential and refrain from donating sperm during participation the study.

Exclusion Criteria:

* Receipt of anticancer therapy or participation in another interventional clinical study within 14 days before the first administration of study drug with the following exceptions: Immunotherapy or biological therapy (eg, monoclonal antibodies) within 21 days the first administration of study drug; 6 weeks for mitomycin-C or nitrosoureas; 7 days for tyrosine kinase inhibitors.
* Radiotherapy within 14 days of first dose of study treatment with the following exceptions: 28 days for pelvic radiotherapy; 6 months for thoracic region radiotherapy that is > 30 Gy.
* Toxicity of prior therapy and/or complications from surgical intervention that has not recovered to ≤ Grade 1 or baseline within 7 days before starting study drug treatment (with the exception of anemia not requiring transfusion support and any grade of alopecia). Note: Endocrinopathy, if well-managed, is not exclusionary and should be discussed with sponsor medical monitor.
* Receipt of prior systemic treatment with an arginase inhibitor
* Immune-related toxicity during prior checkpoint inhibitor therapy for which permanent discontinuation of therapy is recommended (per product label or consensus guidelines), OR any immune-related toxicity requiring intensive or prolonged immunosuppression to manage (with the exception of endocrinopathy that is well controlled on replacement hormones).
* Active autoimmune disease requiring systemic immunosuppression in excess of physiologic maintenance doses of corticosteroids (> 10 mg of prednisone or equivalent).
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Known active hepatitis A virus, hepatitis B virus, or hepatitis C virus infection.
* Known HIV infection.
* Active infections requiring systemic therapy.
* Known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures and/or known hypersensitivity ≥ Grade 3, or severe reaction, to study treatments or any of their excipients or additives.
* Participants with impaired cardiac function or clinically significant cardiac disease.
* Evidence of interstitial lung disease or active, noninfectious pneumonitis or a history of interstitial lung disease.
* Participant is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of treatment-emergent adverse events in participants receiving single-agent INCMGA00012 | Up to approximately 2 years
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 1: Number of treatment-emergent adverse events in participants receiving single-agent INCB001158 | Up to approximately 2 years
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Part 2: Number of treatment-emergent adverse events in participants receiving INCB001158 in combination with INCMGA00012 | Up to approximately 2 years
  Defined as any adverse event either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Part 1: Cmax of single-agent INCMGA000012 | Up to 15 days
  Maximum observed plasma or serum concentration.
Part 1: Cmax of single-agent INCB001158 | Up to 15 days
  Maximum observed plasma or serum concentration.
Part 1: Tmax of single-agent INCMGA000012 | Up to 15 days
  Time to maximum concentration.
Part 1: Tmax of single-agent INCB001158 | Up to 15 days
  Time to maximum concentration.
Part 1: Cmin of single-agent INCMGA000012 | Up to 15 days
  Minimum observed plasma or serum concentration over the dose interval.
Part 1: Cmin of single-agent INCB001158 | Up to 15 days
  Minimum observed plasma or serum concentration over the dose interval.
Part 1: AUCt of single-agent INCMGA000012 | Up to 15 days
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Part 1: AUCt of single-agent INCB001158 | Up to 15 days
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Part 1: t½ of single-agent INCMGA000012 | Up to 15 days
  Apparent terminal-phase disposition half-life.
Part 1: t½ of single-agent INCB001158 | Up to 15 days
  Apparent terminal-phase disposition half-life.
Part 2: Cmax of INCMGA00012 and INCB001158 as a combination treatment | Up to 15 days
  Maximum observed plasma or serum concentration.
Part 2: Tmax of INCMGA00012 and INCB001158 as a combination treatment | Up to 15 days
  Time to maximum concentration.
Part 2: Cmin of INCMGA00012 and INCB001158 as a combination treatment | Up to 15 days
  Minimum observed plasma or serum concentration over the dose interval.
Part 2: AUCt of INCMGA00012 and INCB001158 as a combination treatment | Up to 15 days
  Area under the plasma or serum concentration-time curve from time = 0 to the last measurable concentration at time = t.
Part 2: t½ of INCMGA00012 and INCB001158 as a combination treatment | Up to 15 days
  Apparent terminal-phase disposition half-life.
Part 1 and Part 2: Overall response rate with single-agent INCMGA00012 | Up to 2 years
  Defined as the percentage of participants experiencing a partial response (PR) or complete response (CR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Part 1 and Part 2: Overall response rate with single-agent INCB001158 | Up to 2 years
  Defined as the percentage of participants experiencing a PR or CR as determined by the investigator according to RECIST v1.1.
Part 1 and Part 2: Overall response rate with INCMGA00012 in combination with INCB001158 | Up to 2 years
  Defined as the percentage of participants experiencing a PR or CR as determined by the investigator according to RECIST v1.1.
Part 1 and Part 2: Disease control rate with single-agent INCMGA00012 | Up to 2 years
  Defined as the number of participants maintaining either an overall response rate or stable disease according to RECIST v1.1.
Part 1 and Part 2: Disease control rate with single-agent INCB001158 | Up to 2 years
  Defined as the number of participants maintaining either an overall response rate or stable disease according to RECIST v1.1.
Part 1 and Part 2: Disease control rate with INCMGA00012 in combination with INCB001158 | Up to 2 years
  Defined as the number of participants maintaining either an overall response rate or stable disease according to RECIST v1.1.
Part 1 and Part 2: Duration of response with single-agent INCMGA00012 | Up to 2 years
  Defined as the time from first observed response until onset of disease progression according to RECIST v1.1 or death due to any cause.
Part 1 and Part 2: Duration of response with single-agent INCB001158 | Up to 2 years
  Defined as the time from first observed response until onset of disease progression according to RECIST v1.1 or death due to any cause.
Part 1 and Part 2: Duration of response with INCMGA00012 in combination with INCB001158 | Up to 2 years
  Defined as the time from first observed response until onset of disease progression according to RECIST v1.1 or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Ueda, MD, PhD, MBA, Study Director — Incyte Biosciences Japan GK
Locations (2):
- Japan (2):
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa

IPD SHARING:
Plan to Share IPD: No